CLINICAL TRIAL: NCT04772456
Title: Correlation of Hyperpolarized 13C-pyruvate Metabolic Magnetic Resonance Imaging and Tumor Histopathology in Patients With Infiltrating Gliomas
Brief Title: Hyperpolarized 13C-pyruvate Metabolic MRI With Infiltrating Gliomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Dirk Mayer, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-00086612
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- metabolic MRI (Experimental): Single-arm study in patients who have Glioma Perform metabolic magnetic resonance imaging on patient have a Glioma cancer to understand if metabolic MRI can be safely performed on this population
  Interventions: Drug: Hyperpolarized 13C-Pyruvate

INTERVENTIONS:
Drug: Hyperpolarized 13C-Pyruvate — Hyperpolarized Pyruvate (13C) Injection, containing spin-polarized ("hyperpolarized") [ 13C]pyruvate, is being studied as a diagnostic agent in combination with 13C spectroscopic MR imaging. The aim is to visualize [13C]pyruvate and its metabolites and thereby distinguish between anatomical areas with normal vs. abnormal metabolism, which should be useful in diagnosing and characterizing, for example, malignancy.
  Hyperpolarized Pyruvate (13C) Injection and [13C]pyruvate are general terms used throughout this brochure, that refer to all 13C labeling patterns, such as [1- 13C]pyruvate, [2- 13C]pyruvate and [1,2- 13C]pyruvate. From biological and safety standpoints, pyruvate with each of the labeling patterns behaves identically in the human body [Koletzko et al., 1997].

SUMMARY:
The purpose of this study is to examine the safety and feasibility of performing hyperpolarized metabolic MRI in the diagnosis of brain tumor. This study will also assess the accuracy of hyperpolarized metabolic MRI to diagnose intermediate to patients with infiltrating gliomas and examine the added utility of metabolic MRI over standard MRI imaging

The FDA is allowing the use of hyperpolarized [1-13C] pyruvate (HP 13C-pyruvate) in this study.

Up to 5 patients may take part in this study at the University of Maryland, Baltimore (UMB).

ELIGIBILITY:
Inclusion Criteria:

* • Patients with a new brain lesion interpreted as suspected infiltrating gliomas including but not limited to (diffuse astrocytoma WHO grade 2; oligodendroglioma WHO grade 2 and 3; anaplastic astrocytoma WHO grade 3; astrocytoma WHO grade 4), OR, patients with prior history of infiltrating glioma scheduled for surgery for tumor biopsy or resection.

  * Ages 18-80, including male and female
  * Suitable to undergo contrast-enhanced MRI
  * Negative serum pregnancy test

Exclusion Criteria:

* Inability to undergo MRI scan
* Inability to receive IV contrast secondary to severe reaction or renal insufficiency.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of metabolic MRI to diagnose Glioma | Within three years post treatment
  To study the accuracy of hyperpolarized metabolic MRI to diagnose Glioma Cancer. We will compare the prediction of cancer from the MRI scan compared to actual diagnosis of cancer by any subsequent workup or procedure the participant undergoes. Prediction of cancer from MRI scan will be performed by assigning a standardized score . Actual diagnosis of cancer will be based on tissue pathology.

SECONDARY OUTCOMES:
Utility of metabolic MRI over standard MRI imaging in the diagnosis of Glioma cancer | Within three years post treatment
  To examine the added utility of metabolic MRI over standard MRI imaging. 3. We will quantify the number of participants in which the MRI provided extra information that otherwise was not available during the course of the patient's workup.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Mayer, Dr. rer. nat, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Rosy Njonkou Tchoquessi, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No